CLINICAL TRIAL: NCT04790916
Title: A Double-Blind, Randomized, Parallel-Group, Phase 2 Study to Investigate the Effect of RO7049665 on the Time to Relapse Following Steroid Tapering in Patients With Autoimmune Hepatitis
Brief Title: Effect of RO7049665 on the Time to Relapse Following Steroid Tapering in Participants With Autoimmune Hepatitis (AIH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A lack of efficacy was seen with RO7049665 in a study of ulcerative colitis. This reduces the likelihood that the drug is effective in autoimmune hepatitis.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP42698; 2020-003990-23 (EudraCT Number)
Record Dates: First submitted 2021-03-08; First posted 2021-03-10 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-11

CONDITIONS: Autoimmune Hepatitis; Autoimmune Chronic Hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RO7049665 3.5 mg (Experimental): Participants will receive RO7049665 3.5 mg, administered as subcutaneous (SC) injection, every 2 weeks (Q2W) until participants experience relapse or the study is closed.
  Interventions: Drug: RO7049665
- RO7049665 7.5 mg (Experimental): Participants will receive RO7049665 7.5 mg, administered as SC injection, Q2W until participants experience relapse or the study is closed.
  Interventions: Drug: RO7049665
- Placebo (Placebo Comparator): Participants will receive RO7049665-matching placebo, administered as SC injection, Q2W until participants experience relapse or the study is closed.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RO7049665 — RO7049665, subcutaneous injection, Q2W.
  Arms: RO7049665 3.5 mg; RO7049665 7.5 mg
Other: Placebo — RO7049665-matching placebo, subcutaneous injection, Q2W.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the effect of RO7049665 on time to relapse following forced corticosteroid (CCS) tapering as measured by the hazard ratio between RO7049665 7.5 milligrams (mg) and placebo arm.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a definite diagnosis of AIH (type 1, 2 and 3) as per simplified or revised original diagnostic criteria
* Participants who have been in biochemical remission for > 2 years (or less if according to the local practice) prior to randomization
* Participants who have been on stable treatment (corticosteroids [CCSs] +/- non-specific immunosuppressants [NSIs]) for at least 3 months prior to randomization and who have not had a dose increase in the previous 6 months prior to randomization
* No signs of liver inflammation on a liver biopsy taken no more than 12 months prior to randomization
* Participants with AIH who have previously not attempted (or not attempted in the last 3 years, if this is the local practice) to taper CCSs to 0 mg/day
* Body mass index within the range of 18-35 kilograms per meter square (kg/m^2)
* Women of childbearing potential who agree to remain abstinent or use at least one acceptable contraceptive method during the treatment period and for at least 28 days after the final dose of study drug

Exclusion Criteria:

* Participants with cirrhosis (F4 fibrosis by Fibroscan®) with significant impairment of liver function (Child Pugh category B or C)
* Any other autoimmune disease requiring immunomodulating treatment
* History of infection with hepatitis B, human immunodeficiency virus, active hepatitis C virus (HCV) infection, detection of replicating cytomegalovirus (CMV) or Epstein-Barr virus (EBV)
* Active infections requiring systemic therapy with antibiotic, antiviral, or antifungal treatment or febrile illness within 7 days before Day-1
* History of primary or acquired immunodeficiency
* Pregnant or lactating female participants
* Symptomatic herpes zoster within 3 months prior to screening
* History of active or latent tuberculosis or a positive Quantiferon Gold test
* History of clinically significant severe drug allergies, multiple drug allergies, allergy to any constituent of the product, or intolerance to topical steroids
* Lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years and in situ carcinoma of the cervix that was completely removed surgically. Breast cancer within the past 10 years
* Significant uncontrolled comorbidity, such as cardiac, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders
* Any condition or disease detected during the medical interview/physical examination that would render the participant unsuitable for the study, place the participant at undue risk, or interfere with the ability of the participant to complete the study in the opinion of the Investigator
* CCSs of <5 mg/day, or <2.5 mg CCSs plus immune suppressant, or <3 mg/day budesonide with or without immune suppressant
* CCSs >20 mg/day or >9 mg/day budesonide
* Non-specific immunosuppressant (NSI) daily dose higher than recommended standard of care therapy
* T or B cell-depleting therapy within the last 12 months or T- or B-cell number below normal due to depleting therapy
* Leukocyte apheresis within 12 weeks of screening
* Donation of blood or blood products in excess of 500 milliliters (mL) within 3 months prior to screening.
* Exposure to any investigational treatment within 6 months prior to Day 1
* Abnormal hematologic, hepatic enzyme, hepatic function, or biochemistry values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- The Alfred Hospital - Professor Stuart Roberts' Clinic - The Alfred Centre Location, Melbourne, Victoria, Australia
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Universite de Montreal - Centre Hospitalier de l'Universite de Montreal CHUM - Hopital Saint-Luc, Montreal, Quebec
- Martin Zeitz Centrum für Seltene Erkrankungen ZSE Hamburg, Hamburg, Germany
- Italy (2):
  - IRCCS Saverio De Bellis; Anatomia Patologica, Castellana Grotte, Apulia
  - Ospedale San Gerardo, Monza, Lombardy
- Netherlands (2):
  - Amsterdam UMC - location AMC, Amstermdam
  - Radboud Universiteit - Radboud Universitair Medisch Centrum Radboudumc, Nijmegen
- Centro Hospitalar de Vila Real, Vila Real, Portugal
- South Korea (3):
  - Pusan National University Hospital; division of pulmonology, Busan
  - Korea University Ansan Hospital, Gyeonggi-do
  - University of Ulsan College of Medicine - Asan Medical Center (AMC) - Asan Liver Center, Seoul
- United Kingdom (2):
  - King College Hospital NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Period: Overall Study
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Groups:
- Total: Total of all reporting groups
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male [unit: participants]
Ethnicity (NIH/OMB) [unit: participants]
Race (NIH/OMB) [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse for RO7049665 7.5 mg Versus Placebo
Description: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Time Frame: From randomization (Day 1) up to relapse or end of the study (up to approximately 25 months)
Population: as for baseline characteristics
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change From Baseline in Alanine Aminotransferase (ALT)
Description: as for outcome 1
Time Frame: Up to end of the study (up to approximately 25 months)
Population: as for baseline characteristics
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST)
Description: as for outcome 1
Time Frame: Up to end of the study (up to approximately 25 months)
Population: as for baseline characteristics
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Immunoglobulin G (IgG)
Description: as for outcome 1
Time Frame: Up to end of the study (up to approximately 25 months)
Population: as for baseline characteristics
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Time to Relapse for RO7049665 3.5 mg Versus Placebo
Description: as for outcome 1
Time Frame: From Randomization (Day 1) up to relapse or end of the study (up to approximately 25 months)
Population: as for baseline characteristics
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: as for outcome 1
Time Frame: Up to end of the study (up to approximately 25 months)
Population: as for baseline characteristics
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Emergence and Neutralizing Potential
Description: as for outcome 1
Time Frame: Up to end of the study (up to approximately 25 months)
Population: as for baseline characteristics
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Description: The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.
Arm/Group | RO7049665 3.5 mg | RO7049665 7.5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor. Only 2 participants were enrolled in this study. Based on the low enrollment number, no data is reported here in order to protect and maintain participant privacy/confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT04790916/Prot_SAP_000.pdf